CLINICAL TRIAL: NCT01776788
Title: Effect of Short-Term Intensive Insulin Sequential Exenatide Therapy on β-cell Function and Glycemic Remission Rate in Newly Diagnosed Type 2 Diabetic Patients
Brief Title: Effect of Short-Term Intensive Insulin Sequential Exenatide Therapy in Newly Diagnosed Type 2 Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: bmd-201207-xm
Record Dates: First submitted 2013-01-22; First posted 2013-01-28 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2013-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Lispro; Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- insulin lispro injection, exenatide injection (Experimental)
  Interventions: Drug: insulin lispro injection, exenatide injection
- insulin lispro injection (Active Comparator)
  Interventions: Drug: insulin lispro injection

INTERVENTIONS:
Drug: insulin lispro injection, exenatide injection — First, Patients in the exenatide group will receive short-term continuous subcutaneous insulin (CSII)therapy. The doses will be titrated every day in order to attain the glycaemic goal which is defined as a fasting capillary blood glucose of less than 6.1 mmol/L and capillary blood glucose at 2 h after each of three meals of less than 8.0 mmol/L. Treatments will be maintained for 2 weeks after the glycaemic target will be reached. Then, patients will Sequential be treated with 5 mcg bid for 4 weeks and then 10 mcg bid for 8 weeks. After interventions will be stopped, patients will be instructed to continue diet and physical exercise only and will be followed-up with glycaemic monitoring monthly
  Arms: insulin lispro injection, exenatide injection
Drug: insulin lispro injection — Patients in the control group will receive insulin with an insulin pump. The doses will be titrated every day in order to attain the glycaemic goal. Treatments will be maintained for 2 weeks after the glycaemic target will be reached. Then interventions will be stop, patients will be instructed to continue diet and physical exercise only and will be followed-up with glycaemic monitoring monthly.
  Arms: insulin lispro injection

SUMMARY:
The randomized, controlled trial is to investigate and evaluate the effects of short-term continuous subcutaneous insulin infusion (CSII) sequential exenatide therapy on β-cell function, long-term glycemic control and glycemic remission rate in newly diagnosed type 2 diabetic patients.

DETAILED DESCRIPTION:
The UK Prospective Diabetes Study has shown that β-cell function progressively deteriorates over time in people with type 2 diabetes mellitus, irrespective of lifestyle and existing pharmacological interventions. The progressive nature of type 2 diabetes is one of the major challenges in the treatment of affected patients, and agents that could alter the natural history of this condition would add greatly to current treatment approaches. Short-term intensive insulin therapy of newly diagnosed type 2 diabetes will improve beta-cell function and usually leading to a temporary remission time. The effect of GLP-1 receptor agonists on beta-cells is stimulation of glucose-dependent insulin release, followed by enhancement of insulin biosynthesis. It is stimulating beta-cell proliferation, induction of islet neogenesis, and inhibition of ß-cell apoptosis. Exenatide is synthetic exendin-4, GLP-1 receptor agonist. Exenatide exerts direct effects on β-cell, which indicates that may contribute to delay disease progression. However, no study has evaluated effect of short-term intensive insulin sequential exenatide therapy model on β-cell function and glycemic remission rate in newly diagnosed type 2 diabetic patients. This current study is thus designed to evaluate effect of short-term intensive insulin sequential exenatide therapy model on β-cell function , glycemic control and glycemic remission rate in newly diagnosed type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. newly-diagnosed type 2 diabetic patients, drug naïve
2. age 30~70 years
3. FPG 7.0~16.7mmol/L
4. BMI 20~35 kg/m2, stable body weight (≤10% variation) for at least 3 months prior to screening
5. female patients of reproductive age should practice a reliable method of birth control throughout the study

Exclusion Criteria:

1. acute or severe chronic diabetic complications
2. Recently suffered from MI or CVA.
3. severe gastrointestinal disease
4. other severe intercurrent illness
5. serum aminotransferase (ALT and AST) level higher than 2 times of the upper normal limits and/or serum creatinie≥133µmol/L (1.5mg/dL)
6. tested positive for glutamic acid decarboxylase antibody
7. use of weight loss drugs, corticosteroids, drugs known to affect gastrointestinal motility, transplantation medications, or any investigational drug
8. history of pancreatitis
9. Pregnant or lactation women.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2012-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
the glycemic remission rate in different groups | one year

SECONDARY OUTCOMES:
the improvement of β-cell function in different groups. | one year
the time of glycemic remission in different groups | one year

CONTACTS AND LOCATIONS:
Overall Officials: Xue-jun Li, MD,PhD, Study Director — The First Affiliated Hospital of Xiamen University, China
Locations (1):
- The first afilliated hospital of Xiamen university, Xiamen, Fujian, China